CLINICAL TRIAL: NCT04338945
Title: Impact of Pandemic COVID-19 on Surgical Specialities Residents in Italy: an Italian Polispecialistic Society of Young Surgeons (S.P.I.G.C.) Survey
Brief Title: Impact of Pandemic COVID-19 on Surgical Specialities Residents in Italy
Status: Completed | Type: Observational
Sponsor: Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia (Other)
Responsible Party: Principal Investigator, Simone Ferrero, MD, Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia
Other Study IDs: COVID-ItaliansurgRES-SPIGC
Record Dates: First submitted 2020-04-07; First posted 2020-04-08 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: COVID
Keywords: resident wellness; surgical residency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residents in surgical areas
  Interventions: Behavioral: COVID-surgRES questionaire

INTERVENTIONS:
Behavioral: COVID-surgRES questionaire — The questionaire gives a multidimensional assessment of residents' impression with regard to impact of COVID emergency on Italian specialist training programs

SUMMARY:
The Coronavirus Emergency has severely affected Italian Healthcare National System. This event made it necessary to adopt extraordinary containment measures and to allocate extraordinary resources in Italian hospitals. In many centers routinely elective surgical activity has been decreased or even completely abolished. We believe that this exceptional condition is being consequently having a significant impact on surgical training programs.

DETAILED DESCRIPTION:
Purpose of this investigation, organized by the Italian Polispecialistic Society of Young Surgeons (S.P.I.G.C.), is to establish the impact of COVID-19 emergency in the work and training activities of Italian surgical residents.

There will be collected the residents' impressions by completing a survey on this topic. A sub-analysis for each pandemic wave (first, second, third) will be done.

ELIGIBILITY:
Inclusion Criteria:

- Residents in the following surgical specialities: cardiothoracic surgery, colon and rectal surgery, general surgery, gynecology and obstetrics, gynecologic oncology, neurological surgery, ophthalmic surgery, oral and maxillofacial surgery, orthopaedic surgery, otorhinolaryngology, pediatric surgery, plastic and maxillofacial surgery, urology, and vascular surgery

Exclusion Criteria:

* Undergratuated and postgraduated students
* Consultants in surgical areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Italian medical residents in surgical areas
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Measure of the impact of first wave of COVID Pandemic on surgical specialist training programs | 1-3 months after the beginning of COVID emergency in Italy
  Analysis of this outcome with regard to the different surgical subspecialities and different Italian medical centers
Measure of the impact of second wave of COVID Pandemic on surgical specialist training programs | 1 year after the beginning of COVID emergency in Italy
  Analysis of this outcome with regard to the different surgical subspecialities and different Italian medical centers
Measure of the impact of third wave of COVID Pandemic on surgical specialist training programs | 2 years after the beginning of COVID emergency in Italy
  Analysis of this outcome with regard to the different surgical subspecialities and different Italian medical centers

SECONDARY OUTCOMES:
Measure of impact of first wave of COVID Pandemic on wellness of residents | 1-3 months after the beginning of COVID emergency in Italy
  Analysis of this outcome with regard to the different surgical subspecialities and different Italian medical centers
Measure of impact of second wave of COVID Pandemic on wellness of residents | 1 year after the beginning of COVID emergency in Italy
  Analysis of this outcome with regard to the different surgical subspecialities and different Italian medical centers
Measure of impact of third wave of COVID Pandemic on wellness of residents | 2 years after the beginning of COVID emergency in Italy
  Analysis of this outcome with regard to the different surgical subspecialities and different Italian medical centers

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - U.O.C. Chirurgia Generale Universitaria "V. Bonomo", Bari
  - Ospedale Perrino Asl Brindisi, Brindisi
  - Dipartimento di scienze mediche e chirurgiche, Università di Catanzaro, Catanzaro
  - Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - IRCCS Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale Cristo re, Roma